CLINICAL TRIAL: NCT00046293
Title: ReoPro Retavase Reperfusion of Stroke Safety Study-Imaging Evaluation With Computed Tomography (ROSIE-CT)
Brief Title: ReoPro and Retavase to Treat Acute Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Steven J. Warach, M.D./National Institute of Neurological Disorders and Stroke, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020301; 02-N-0301
Record Dates: First submitted 2002-09-25; First posted 2002-09-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-08

CONDITIONS: Cerebrovascular Accident
Keywords: Stroke; Abciximab; Retavase; MRI; Cerebral Blood Flow
MeSH Terms: conditions — Stroke | interventions — Abciximab

INTERVENTIONS:
Drug: Reopro
Drug: Retrovase

SUMMARY:
This study will determine the dose of Retavase that can safely be combined with ReoPro in treating acute ischemic stroke (stroke resulting from a blood clot in the brain). ReoPro and Retavase are currently approved by the Food and Drug Administration to treat heart problems caused by blockage of heart arteries. The only therapy approved by the Food and Drug Administration to treat ischemic stroke is the clot buster drug rt-PA. This treatment is effective only if begun within 3 hours of onset of the stroke, however, and most patients do not get to the hospital early enough to benefit from it.

Patients between 18 and 80 years of age who have had a mild or moderate acute stroke between 3 and 24 hours before starting study drugs may be eligible for this study. Candidates will be screened with a medical history and physical examination, blood tests, rating of neurological deficits such as cognition deficits or problems walking that resulted from the stroke, and a computed tomography (CT) scan of the head. CT involves the use of specialized X-rays to obtain images of the brain. The patient lies on a table that is moved into a cylindrical machine (the scanner) for the imaging study, which usually takes about 5 to 10 minutes.

All participants will receive 0.25 mg/kg of ReoPro (maximum dose of 30 mg). The drug is infused into the vein over 12 hours. Some patients will also receive one of four doses of Retavase, which may boost the effectiveness of ReoPro in opening the blocked blood vessel. Retavase is given through a needle in the vein over 2 minutes. Patients will be monitored daily until discharge from the hospital, or until day 5, whichever is earlier. Assessments will include physical examinations, blood tests to examine factors involved in blood clotting, and CT scans to evaluate both the response to treatment and drug side effects. They will return for a follow-up examination and CT scan 30 days after treatment.

...

DETAILED DESCRIPTION:
Objectives: This is the companion protocol to the ROSIE protocol. This clinical trial will determine an acceptable dose of reteplase in combination with a fixed dose of abciximab for ischemic stroke 3-24 hours from onset in patients screened with brain CT rather than MRI (as required by the ROSIE protocol). The importance of this study relative to ROSIE will be its relevance to the large proportion of acute stroke patients who cannot have a screening MRI, because of contraindications or unavailability of emergency MRI at their hospital.

Study Population: Patients will be selected by criteria to minimize likelihood of toxicity and maximize likelihood of response. These criteria include age 18-80 years old, patients who cannot get acute MRI because of contraindication to or unavailability of MRI, acute ischemic stroke of moderate severity (NIH Stroke Scale less than or equal to 16 and ischemic changes on CT scan less than approximately one third of the volume of the middle cerebral artery territory), no evidence of hemorrhage on CT, and no other clinical, radiological or laboratory features associated with increased risk of hemorrhage with thrombolytic therapy.

Design: The study is open-label, dose escalation, safety and proof of principle study of the combination of intravenous abciximab and reteplase. A fixed dose of abciximab will be used in all patients: 0.25 mg/kg bolus (to a maximum of 30 mg) followed by a 0.125 microgram/kg/minute infusion (to a maximum of 10.0 microgram/minute) for 12 hours. The five dosing groups for the reteplase dose are 0U, 2.5 U, 5.0 U, 7.5 U, and 10.0 U. A maximum of 72 patients will be treated using an adaptive statistical design. Non-investigation patient management will be standardized across all patients according to the NIH Stroke Center Clinical Care Pathway.

Outcome Measures: The primary efficacy endpoint for response will be clinical improvement (complete recovery or improvement of 4 points or more on the NIH Stroke Scale) at 24 hours after start of therapy. The primary safety endpoint for determination of toxicity will be any one of the following: symptomatic intracranial hemorrhage (ICH), major systemic hemorrhage, or other serious adverse event related to study drug administration, including death, within 48 hours from start of therapy. The maximum acceptable rate of toxicity will be 10% of patients treated at any dose level and the minimum acceptable rate of response will be 50% of patients at any dose level. The outcomes will be monitored by a Data and Safety Monitoring Committee, which will have the authority to stop or recommend modifications of the trial for safety concerns. Other clinical outcome variables and imaging variables will be recorded and analyzed in secondary and exploratory analyses. If an acceptable dose is identified, then that will be investigated in a subsequent randomized placebo-controlled trial.

ELIGIBILITY:
* INCLUSION CRITERIA

Patients may be enrolled in the study only if they meet all of the following criteria:

Diagnosis of acute ischemic stroke with onset between 3 and 24 hours prior to planned start of study drugs. Acute ischemic stroke is defined as a measurable neurological deficit of sudden onset, presumed secondary to focal cerebral ischemia, and not otherwise attributable to ICH or another disease process. Stroke onset will be defined as the time the patient was last known to be without the new clinical deficit. Patients whose deficits have worsened in the last 24 hours are not eligible if their first symptoms started more than 24 hours before. If the stroke started during sleep, stroke onset will be recorded as the time the patient was last known to be intact. A careful history is important to determine when the patient was last without the presenting deficits.

Disabling neurological deficit attributable to the acute stroke at the start of study drugs.

NIHSS less than or equal to16

Age 18 - 80 years, inclusive.

Patients not evaluable for the ROSIE protocol because of MRI contraindication or MRI unavailability or technically inadequate diffusion and perfusion MRI.

EXCLUSION CRITERIA

Patients will be excluded from the study for any of the following reasons:

General

Current participation in another study with an investigational drug or device within, prior participation in the present study, or planned participation in another therapeutic trial, prior to the final assessment in this trial.

Time interval since stroke onset of less than 24 hours is impossible to determine with high degree of confidence.

Symptoms suggestive of subarachnoid hemorrhage, even if CT scan is negative for hemorrhage.

Evidence of acute myocardial infarction defined as having at least two of the following three features: 1) Chest pain suggestive of cardiac ischemia 2) EKG findings of ST elevation of more greater than 0.2 mV in 2 contiguous leads, new onset left bundle branch block, ST segment depression, or T-wave inversion 3) Elevated troponin I

Women known to be pregnant, lactating or having a positive or indeterminate pregnancy test.

Patients who would refuse blood transfusions if medically indicated

Stroke Related

Neurological deficit that has led to stupor or coma (NIHSS level of consciousness score greater than or equal to 2).

High clinical suspicion of septic embolus.

Minor stroke with non-disabling deficit or rapidly improving neurological symptoms.

Baseline NIHSS greater than 16.

MRI/CT Related

Evidence of acute or chronic ICH by head CT.

CT evidence of non-vascular cause for the neurological symptoms.

Signs of mass effect causing shift of midline structures.

Patient excluded from the ROSIE protocol by MRI findings.

Acute ischemic changes on CT larger than approximately one third of the territory of the middle cerebral artery territory by qualitative assessment.

Safety Related

Persistent hypertension with systolic BP greater than 185 mmHg or diastolic BP greater than 110 mmHg (mean of 3 consecutive arm cuff readings over 20-30 minutes), not controlled by antihypertensive therapy or requiring nitroprusside for control.

Anticipated need for major surgery within 72 hours after start of study drugs, e.g., carotid endarterectomy, hip fracture repair.

Any intracranial surgery, serious head trauma (any head injury that required hospitalization), or stroke within the past 3 months.

Stroke within the past 3 months.

History of ICH at any time in the past.

Major trauma at the time of stroke, e.g., hip fracture.

Blood glucose greater than 200 mg/dl.

Presence or history of intracranial neoplasm or arteriovenous malformation.

Intracranial aneurysm, unless surgically treated greater than 3 months.

Major hemorrhage in past 21 days.

Major surgery, serious trauma, lumbar puncture, arterial puncture at a non-compressible site, or biopsy of a parenchymal organ in last 14 days. Major surgical procedures include but are not limited to the following: major thoracic or abdominopelvic surgery, neurosurgery, major limb surgery, carotid endarterectomy or other vascular surgery, and organ transplant. For non-listed procedures, the operating surgeon should be consulted to assess the risk.

Presumed or documented history of vasculitis.

Known systemic bleeding disorder, e.g., von Willebrand's disease, hemophilia, others.

Platelet count less than 100,000 cells/mL.

Congenital or acquired coagulopathy (e.g., secondary to anticoagulants) causing either of the following:

1. Activated partial thromboplastin time (aPTT) prolongation greater than 2 seconds above the upper limit of normal for local laboratory, except if due to isolated factor XII deficiency. Protamine sulfate reversal of heparin effect does not alleviate this criterion.
2. INR greater than or equal to 1.4. Patients receiving warfarin prior to entry are eligible provided INR is less than 1.4 and warfarin can be safely discontinued for at least 48 hours.

Potentially Interfering with Outcome Assessment

Life expectancy less than 3 months.

Other serious illness, e.g., severe hepatic, cardiac, or renal failure; acute myocardial infarction; or a complex disease that may confound treatment assessment.

Serum creatinine, AST or ALT greater than 3 times the upper limit of normal for the local laboratory.

Drug Related

Treatment of the qualifying stroke with any thrombolytic or GPIIbIIIa inhibitor outside of this protocol.

Any administration of a thrombolytic drug in the prior 7 days.

Treatment of the qualifying stroke with intravenous heparin unless aPTT prolongation is no greater than 2 seconds above the upper limit of normal for local laboratory prior to study drug initiation.

Treatment of the qualifying stroke with a low molecular weight heparinoid.

Previous administration of abciximab, if known.

Known allergy to murine proteins.

Anticoagulation caused by herbal therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2002-09-24; Primary Completion 2007-07-20 (Actual); Study Completion 2007-07-20 (Actual)

PRIMARY OUTCOMES:
Clinical improvement at 24 hours after start of therapy.

SECONDARY OUTCOMES:
Final infarct volume at day 30 CT adjusted for patient age and baseline NIHSS.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. Tissue plasminogen activator for acute ischemic stroke. N Engl J Med. 1995 Dec 14;333(24):1581-7. doi: 10.1056/NEJM199512143332401. PMID 7477192
- [Background] Hacke W, Kaste M, Fieschi C, von Kummer R, Davalos A, Meier D, Larrue V, Bluhmki E, Davis S, Donnan G, Schneider D, Diez-Tejedor E, Trouillas P. Randomised double-blind placebo-controlled trial of thrombolytic therapy with intravenous alteplase in acute ischaemic stroke (ECASS II). Second European-Australasian Acute Stroke Study Investigators. Lancet. 1998 Oct 17;352(9136):1245-51. doi: 10.1016/s0140-6736(98)08020-9. PMID 9788453
- [Background] Hacke W, Kaste M, Fieschi C, Toni D, Lesaffre E, von Kummer R, Boysen G, Bluhmki E, Hoxter G, Mahagne MH, et al. Intravenous thrombolysis with recombinant tissue plasminogen activator for acute hemispheric stroke. The European Cooperative Acute Stroke Study (ECASS). JAMA. 1995 Oct 4;274(13):1017-25. PMID 7563451